CLINICAL TRIAL: NCT02404480
Title: A Phase 1 Study of PTC596 in Patients With Advanced Solid Tumors
Brief Title: PTC596 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTC596-ONC-001-AST
Record Dates: First submitted 2015-03-24; First posted 2015-03-31 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — PTC596

STUDY DESIGN:
Intervention Model Description: Open-label, first-in-human, safety and pharmacokinetic (PK)
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1 (Experimental): PTC 596 administered twice daily- Dose level 0.65mg/kg
  Interventions: Drug: PTC596
- Cohort 2 (Experimental): PTC 596 administered twice daily-Dose level 1.3mg/kg
  Interventions: Drug: PTC596
- Cohort 3 (Experimental): PTC 596 administered twice daily-2.6mg/kg
  Interventions: Drug: PTC596
- Cohort 4 (Experimental): PTC 596 administered twice daily-Dose level 5.2mg/kg
  Interventions: Drug: PTC596
- Cohort 5 (Experimental): PTC 596 administered twice daily-Dose level 10mg/kg
  Interventions: Drug: PTC596
- Cohort 6 (Experimental): PTC 596 administered twice daily-Dose level 7mg/kg
  Interventions: Drug: PTC596
- Cohort 7 (Bio Marker cohort) (Experimental): PTC 596 administered twice daily-Dose level 5.2mg/kg
  Interventions: Drug: PTC596

INTERVENTIONS:
Drug: PTC596 — PTC 596 will be administered orally twice a day until unmanageable toxicity, disease progression, or withdrawal of consent is noted

SUMMARY:
This is a Phase 1, open-label, first-in-human, safety and pharmacokinetic study of PTC596 in patients with advanced cancer.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, first-in-human, safety and pharmacokinetic (PK) study of PTC596 in patients with advanced cancer. A variation of the traditional 3+3 dose escalation design will be employed.

PTC596 will be administered orally on a twice a week (biw) schedule. Each 4-week period of drug administration will be considered one cycle. The objective of the study will be to determine the recommended Phase 2 dose (RP2D) and to determine preliminary proof of mechanism of action.

Collectively, data from the Good Laboratory Practice (GLP) and non-GLP studies indicate that 40 mg/kg biw is approximately the severely toxic dose in 10% of animals (STD 10). Therefore, the starting dose in this study will be calculated as one-tenth of the human equivalent dose (HED) of 40 mg/kg biw in rats, which is 0.65 mg/kg biw.

In this study, escalating dose levels will be evaluated to determine the RP2D. Three patients will be enrolled at the starting dose level (0.65 mg/kg biw); if 1 of the 3 patients experiences a dose-limiting toxicity (DLT), an additional 3 patients will be enrolled at the same dose level. Thus, 3 to 6 patients will receive the starting dose level of 0.65 mg/kg. Dose escalation will continue until the occurrence of DLT in ≥2/6 patients at a given dose level. Dose escalation will occur in approximately 100% increments until Grade ≥2, first-cycle toxicity is seen in at least 2 patients across all dose levels, after which dose escalation will occur in smaller (50% or 33%) increments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed solid malignancy that is metastatic or unresectable, for which standard curative measures do not exist, that has progressed on at least one line of standard therapy or for which no standard therapies exists
* Discontinuation of all other therapies (including other investigational drugs, radiotherapy, or chemotherapy) for the treatment of cancer ≥4 weeks (≥6 weeks if nitrosoureas, ≥12 weeks if radiotherapy) before initiation of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* A measured or estimated creatinine clearance (CrCl) ≥60 mL/min/1.73 m2

Exclusion Criteria:

* Prior bone marrow/hematopoietic stem cell transplantation
* History of solid organ, bone marrow, or progenitor cell transplantation
* History of major surgical procedure within 28 days prior to start of study treatment
* Evidence of ongoing systemic bacterial, fungal, or viral infection. Known human immunodeficiency virus (HIV) infection or acquired-immunodeficiency syndrome (AIDS)-related illness
* Any of the following in the past 6 months: myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, congestive heart failure (New York Heart Association Class III or IV), cerebrovascular accident, transient ischemic attack, other arterial thromboembolic event, or pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities | 28 days
  Determine the RP2D based on occurrence of DLTs and/or biological efficacy as determined by biomarker changes.

SECONDARY OUTCOMES:
Adverse effects | 28days
  Define and describe the adverse effects of PTC596 in humans when orally administered on a biw schedule.
Time to Maximum Plasma Concentration (T max) | 28days
  Evaluate the Time to Maximum Plasma Concentration (T max) of PTC596 in humans.
Antitumor activity | 28days
  Describe any preliminary evidence of antitumor activity of PTC596.
Maximum Plasma Concentration (C max) | 28 days
  Evaluate the Maximum Plasma Concentration (C max) of PTC596 in humans
Plasma Concentration at 24 hours | 28days
  Evaluate the Plasma Concentration at 24 hours of PTC596 in humans
Area under the plasma concentration-time curve (AUC) | 28 days
  Evaluate the area under the plasma concentration-time curve (AUC) of PTC 596 in humans.
Terminal half-life (t1/2). | 28 days.
  Evaluate the terminal half-life (t1/2) of PTC 596 in humans.

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — PTC Therapeutics
Locations (4):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Abdouh M, Facchino S, Chatoo W, Balasingam V, Ferreira J, Bernier G. BMI1 sustains human glioblastoma multiforme stem cell renewal. J Neurosci. 2009 Jul 15;29(28):8884-96. doi: 10.1523/JNEUROSCI.0968-09.2009. PMID 19605626
- [Background] American Society of Clinical Oncology; Kris MG, Hesketh PJ, Somerfield MR, Feyer P, Clark-Snow R, Koeller JM, Morrow GR, Chinnery LW, Chesney MJ, Gralla RJ, Grunberg SM. American Society of Clinical Oncology guideline for antiemetics in oncology: update 2006. J Clin Oncol. 2006 Jun 20;24(18):2932-47. doi: 10.1200/JCO.2006.06.9591. Epub 2006 May 22. PMID 16717289
- [Background] Beck B, Blanpain C. Unravelling cancer stem cell potential. Nat Rev Cancer. 2013 Oct;13(10):727-38. doi: 10.1038/nrc3597. PMID 24060864
- [Background] Cao R, Tsukada Y, Zhang Y. Role of Bmi-1 and Ring1A in H2A ubiquitylation and Hox gene silencing. Mol Cell. 2005 Dec 22;20(6):845-54. doi: 10.1016/j.molcel.2005.12.002. PMID 16359901
- [Background] Chiba T, Miyagi S, Saraya A, Aoki R, Seki A, Morita Y, Yonemitsu Y, Yokosuka O, Taniguchi H, Nakauchi H, Iwama A. The polycomb gene product BMI1 contributes to the maintenance of tumor-initiating side population cells in hepatocellular carcinoma. Cancer Res. 2008 Oct 1;68(19):7742-9. doi: 10.1158/0008-5472.CAN-07-5882. PMID 18829528
- [Background] Cho JH, Dimri M, Dimri GP. A positive feedback loop regulates the expression of polycomb group protein BMI1 via WNT signaling pathway. J Biol Chem. 2013 Feb 1;288(5):3406-18. doi: 10.1074/jbc.M112.422931. Epub 2012 Dec 13. PMID 23239878
- [Background] Costa DB, Li S, Kocher O, Feins RH, Keller SM, Schiller JH, Johnson DH, Tenen DG, Halmos B. Immunohistochemical analysis of C/EBPalpha in non-small cell lung cancer reveals frequent down-regulation in stage II and IIIA tumors: a correlative study of E3590. Lung Cancer. 2007 Apr;56(1):97-103. doi: 10.1016/j.lungcan.2006.11.023. Epub 2007 Jan 18. PMID 17239984
- [Background] Douglas D, Hsu JH, Hung L, Cooper A, Abdueva D, van Doorninck J, Peng G, Shimada H, Triche TJ, Lawlor ER. BMI-1 promotes ewing sarcoma tumorigenicity independent of CDKN2A repression. Cancer Res. 2008 Aug 15;68(16):6507-15. doi: 10.1158/0008-5472.CAN-07-6152. PMID 18701473
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Facchino S, Abdouh M, Chatoo W, Bernier G. BMI1 confers radioresistance to normal and cancerous neural stem cells through recruitment of the DNA damage response machinery. J Neurosci. 2010 Jul 28;30(30):10096-111. doi: 10.1523/JNEUROSCI.1634-10.2010. PMID 20668194
- [Background] Fan C, He L, Kapoor A, Rybak AP, De Melo J, Cutz JC, Tang D. PTEN inhibits BMI1 function independently of its phosphatase activity. Mol Cancer. 2009 Nov 10;8:98. doi: 10.1186/1476-4598-8-98. PMID 19903340
- [Background] Glinsky GV, Berezovska O, Glinskii AB. Microarray analysis identifies a death-from-cancer signature predicting therapy failure in patients with multiple types of cancer. J Clin Invest. 2005 Jun;115(6):1503-21. doi: 10.1172/JCI23412. PMID 15931389
- [Background] Guney I, Wu S, Sedivy JM. Reduced c-Myc signaling triggers telomere-independent senescence by regulating Bmi-1 and p16(INK4a). Proc Natl Acad Sci U S A. 2006 Mar 7;103(10):3645-50. doi: 10.1073/pnas.0600069103. Epub 2006 Feb 28. PMID 16537449
- [Background] Kreso A, van Galen P, Pedley NM, Lima-Fernandes E, Frelin C, Davis T, Cao L, Baiazitov R, Du W, Sydorenko N, Moon YC, Gibson L, Wang Y, Leung C, Iscove NN, Arrowsmith CH, Szentgyorgyi E, Gallinger S, Dick JE, O'Brien CA. Self-renewal as a therapeutic target in human colorectal cancer. Nat Med. 2014 Jan;20(1):29-36. doi: 10.1038/nm.3418. Epub 2013 Dec 1. PMID 24292392
- [Background] Li DW, Tang HM, Fan JW, Yan DW, Zhou CZ, Li SX, Wang XL, Peng ZH. Expression level of Bmi-1 oncoprotein is associated with progression and prognosis in colon cancer. J Cancer Res Clin Oncol. 2010 Jul;136(7):997-1006. doi: 10.1007/s00432-009-0745-7. Epub 2009 Dec 19. PMID 20024662
- [Background] Liu L, Andrews LG, Tollefsbol TO. Loss of the human polycomb group protein BMI1 promotes cancer-specific cell death. Oncogene. 2006 Jul 20;25(31):4370-5. doi: 10.1038/sj.onc.1209454. Epub 2006 Feb 27. PMID 16501599
- [Background] Molofsky AV, Pardal R, Iwashita T, Park IK, Clarke MF, Morrison SJ. Bmi-1 dependence distinguishes neural stem cell self-renewal from progenitor proliferation. Nature. 2003 Oct 30;425(6961):962-7. doi: 10.1038/nature02060. Epub 2003 Oct 22. PMID 14574365
- [Background] Nacerddine K, Beaudry JB, Ginjala V, Westerman B, Mattiroli F, Song JY, van der Poel H, Ponz OB, Pritchard C, Cornelissen-Steijger P, Zevenhoven J, Tanger E, Sixma TK, Ganesan S, van Lohuizen M. Akt-mediated phosphorylation of Bmi1 modulates its oncogenic potential, E3 ligase activity, and DNA damage repair activity in mouse prostate cancer. J Clin Invest. 2012 May;122(5):1920-32. doi: 10.1172/JCI57477. Epub 2012 Apr 16. PMID 22505453
- [Background] Nachimuthu S, Assar MD, Schussler JM. Drug-induced QT interval prolongation: mechanisms and clinical management. Ther Adv Drug Saf. 2012 Oct;3(5):241-53. doi: 10.1177/2042098612454283. PMID 25083239
- [Background] Nakamura S, Oshima M, Yuan J, Saraya A, Miyagi S, Konuma T, Yamazaki S, Osawa M, Nakauchi H, Koseki H, Iwama A. Bmi1 confers resistance to oxidative stress on hematopoietic stem cells. PLoS One. 2012;7(5):e36209. doi: 10.1371/journal.pone.0036209. Epub 2012 May 11. PMID 22606246
- [Background] O'Connor ML, Xiang D, Shigdar S, Macdonald J, Li Y, Wang T, Pu C, Wang Z, Qiao L, Duan W. Cancer stem cells: A contentious hypothesis now moving forward. Cancer Lett. 2014 Mar 28;344(2):180-7. doi: 10.1016/j.canlet.2013.11.012. Epub 2013 Dec 11. PMID 24333726
- [Background] Pan MR, Peng G, Hung WC, Lin SY. Monoubiquitination of H2AX protein regulates DNA damage response signaling. J Biol Chem. 2011 Aug 12;286(32):28599-607. doi: 10.1074/jbc.M111.256297. Epub 2011 Jun 15. PMID 21676867
- [Background] Park IK, Qian D, Kiel M, Becker MW, Pihalja M, Weissman IL, Morrison SJ, Clarke MF. Bmi-1 is required for maintenance of adult self-renewing haematopoietic stem cells. Nature. 2003 May 15;423(6937):302-5. doi: 10.1038/nature01587. Epub 2003 Apr 20. PMID 12714971
- [Background] Park IK, Morrison SJ, Clarke MF. Bmi1, stem cells, and senescence regulation. J Clin Invest. 2004 Jan;113(2):175-9. doi: 10.1172/JCI20800. PMID 14722607
- [Background] Siddique HR, Parray A, Tarapore RS, Wang L, Mukhtar H, Karnes RJ, Deng Y, Konety BR, Saleem M. BMI1 polycomb group protein acts as a master switch for growth and death of tumor cells: regulates TCF4-transcriptional factor-induced BCL2 signaling. PLoS One. 2013 May 6;8(5):e60664. doi: 10.1371/journal.pone.0060664. Print 2013. PMID 23671559
- [Background] Silva J, Garcia JM, Pena C, Garcia V, Dominguez G, Suarez D, Camacho FI, Espinosa R, Provencio M, Espana P, Bonilla F. Implication of polycomb members Bmi-1, Mel-18, and Hpc-2 in the regulation of p16INK4a, p14ARF, h-TERT, and c-Myc expression in primary breast carcinomas. Clin Cancer Res. 2006 Dec 1;12(23):6929-36. doi: 10.1158/1078-0432.CCR-06-0788. PMID 17145810
- [Background] Sparmann A, van Lohuizen M. Polycomb silencers control cell fate, development and cancer. Nat Rev Cancer. 2006 Nov;6(11):846-56. doi: 10.1038/nrc1991. PMID 17060944
- [Background] Vrzalikova K, Skarda J, Ehrmann J, Murray PG, Fridman E, Kopolovic J, Knizetova P, Hajduch M, Klein J, Kolek V, Radova L, Kolar Z. Prognostic value of Bmi-1 oncoprotein expression in NSCLC patients: a tissue microarray study. J Cancer Res Clin Oncol. 2008 Sep;134(9):1037-42. doi: 10.1007/s00432-008-0361-y. Epub 2008 Feb 9. PMID 18264721
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- [Background] Wu Z, Min L, Chen D, Hao D, Duan Y, Qiu G, Wang Y. Overexpression of BMI-1 promotes cell growth and resistance to cisplatin treatment in osteosarcoma. PLoS One. 2011 Feb 2;6(2):e14648. doi: 10.1371/journal.pone.0014648. PMID 21311599
- [Background] Wu X, Liu X, Sengupta J, Bu Y, Yi F, Wang C, Shi Y, Zhu Y, Jiao Q, Song F. Silencing of Bmi-1 gene by RNA interference enhances sensitivity to doxorubicin in breast cancer cells. Indian J Exp Biol. 2011 Feb;49(2):105-12. PMID 21428211
- [Background] Zhang P, Iwasaki-Arai J, Iwasaki H, Fenyus ML, Dayaram T, Owens BM, Shigematsu H, Levantini E, Huettner CS, Lekstrom-Himes JA, Akashi K, Tenen DG. Enhancement of hematopoietic stem cell repopulating capacity and self-renewal in the absence of the transcription factor C/EBP alpha. Immunity. 2004 Dec;21(6):853-63. doi: 10.1016/j.immuni.2004.11.006. PMID 15589173
- [Background] Zhang R, Xu LB, Yue XJ, Yu XH, Wang J, Liu C. Bmi1 gene silencing inhibits the proliferation and invasiveness of human hepatocellular carcinoma cells and increases their sensitivity to 5-fluorouracil. Oncol Rep. 2013 Mar;29(3):967-74. doi: 10.3892/or.2012.2189. Epub 2012 Dec 14. PMID 23242307
- [Derived] Yong KJ, Basseres DS, Welner RS, Zhang WC, Yang H, Yan B, Alberich-Jorda M, Zhang J, de Figueiredo-Pontes LL, Battelli C, Hetherington CJ, Ye M, Zhang H, Maroni G, O'Brien K, Magli MC, Borczuk AC, Varticovski L, Kocher O, Zhang P, Moon YC, Sydorenko N, Cao L, Davis TW, Thakkar BM, Soo RA, Iwama A, Lim B, Halmos B, Neuberg D, Tenen DG, Levantini E. Targeted BMI1 inhibition impairs tumor growth in lung adenocarcinomas with low CEBPalpha expression. Sci Transl Med. 2016 Aug 3;8(350):350ra104. doi: 10.1126/scitranslmed.aad6066. PMID 27488898
- See also: Characterization and Chromosomal localization of the human proto-oncogene — http://www.nature.com/articles/6691791
- See also: Human protein atlas — http://www.proteinatlas.org/ENSG00000168283-BMI1/tissue
- See also: Exploratory assessment of dose proportionality — https://www.researchgate.net/publication/5465319_Exploratory_assessment_of_dose_proportionality_Review_of_current_approaches_and_proposal_for_a_practical_criterion
- See also: Dose escalation study design example — https://prsinfo.clinicaltrials.gov/trainTrainer/Dose-Escalation-Design-Fiction-Manuscript.pdf
- See also: Increased polycomb-group oncogene BMI-1expression coorelates with poor prognosis in Hepatocellular carcinoma — https://rd.springer.com/article/10.1007/s00432-007-0316-8?no-access=true